CLINICAL TRIAL: NCT01133262
Title: Effectiveness in Head and Neck Cancer Detection Using PET Insert Device
Brief Title: Effectiveness in Head and Neck Cancer Detection Using Positron Emission Tomography (PET) Insert Device
Status: Withdrawn | Type: Observational
Why Stopped: Feasibility/pilot study of 5 subjects registration not required
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: WashU-Tai10
Record Dates: First submitted 2010-05-26; First posted 2010-05-28 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
We have developed a prototype PET insert device that can be integrated into a clinical PET/computed tomography (CT) scanner to improve its image resolution to approximately 2.5 mm in all 3 dimensions within a reduced imaging field of view (FOV). This zoom-in imaging capability provides 6-fold improvement in volumetric image resolution over the current state-of-the-art clinical PET scanner, offering a tremendous opportunity for cancer imaging applications, in particular for those cases where a lymph node involvement will drastically alter the patient management plan. Accurate diagnosis and staging of head-and-neck cancer is known to be challenging because of the complex anatomy and large number of lymph nodes involved in this region. As a result, head and neck cancer imaging is an ideal candidate for evaluating the clinical usefulness of this novel imaging device.

DETAILED DESCRIPTION:
In this project, we propose to conduct an exploratory clinical trial to investigate the effectiveness of this novel imaging device in detecting small lesions and lymph node involvements in the head and neck region, and compare its results to those obtained from a clinical PET/CT scanner. More specifically, we propose to (1) recruit 5 patients who have confirmed head and neck cancer and are scheduled to receive a whole-body PET/CT scan followed by surgical operation to remove the primary tumor and the regional lymph nodes. These patients will be imaged by a state-of-the-art PET/CT scanner using the standard whole-body PET/CT imaging protocol as standard of care for initial staging. On another day, following consent to participate in this research protocol, A patient will undergo images of the head and neck region using the same type scanner with and without our novel PET insert device attached; (2) The images obtained from the PET insert device will be reviewed by experienced nuclear medicine physicians to identify the extent of lymph node involvement. The PET insert images will be compared to the standard clinical PET/CT images. A detailed image obtained for purposes of research, centered at the level of the head and neck, acquired for approximately 3 times the length of time the standard clinical image is obtained for will also be compared to the PET insert image. Images will also be compared to the pathology report of the surgically removed specimen. (3) Estimate the performance of lesion detection for different sizes of tumors using the standard PET/CT scanner as well as the PET insert device.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically or cytologically confirmed squamous cell carcinoma of the head and neck with suspected lymph node metastasis. Subjects with histological confirmation of squamous cell carcinoma from a lymph node biopsy in the head and neck region for carcinoma of unknown primary would also be eligible.
2. Patient must be scheduled to receive (or have already received) clinical whole body PET/CT scan from a Siemens Biograph 40 PET/CT scanner as their standard of care staging.
3. Patient must be scheduled to receive surgical removal of the primary tumor and the regional lymph nodes. It is preferred that the surgery will occur within 21 days of research PET imaging.
4. Age >18 years, as head and neck cancer is extremely rare in children.
5. Ability of the patient (or legally authorized representative if applicable) to understand and the willingness to sign a written informed consent document.
6. Not currently pregnant or nursing: Female subjects must be either surgically sterile (has had a documented bilateral oophorectomy and/or documented hysterectomy), or post menopausal (cessation of menses for more than 1 year). If of childbearing potential, a urine pregnancy test must be performed within the 24 hour period immediately prior to administration of 18FDG and determined to be negative

Exclusion Criteria:

1. The subject weight will be limited to 250 lbs and below due to the size limitations of the prototype PET insert device.
2. Subjects who are claustrophobic
3. Subjects with poorly controlled diabetes (fasting blood glucose >200mg/dL)
4. Subjects with prior head/neck surgery or radiation as this may disturb the natural architecture of the tissues and impede the imaging analysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with biopsy proven squamous cell carcinoma of the head and neck with suspected lymph node metastasis
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-06; Study Completion 2011-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Yuan-Chuan Tai, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Barnes-Jewish Hospital, St Louis, Missouri, United States

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu